CLINICAL TRIAL: NCT06825611
Title: Detecting and Monitoring Scoliosis Without Radiography: Standard Radiographic Monitoring Program Versus Self-Screening with Momentum SpineTM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Momentum Health Inc. (Industry)
Responsible Party: Principal Investigator, Lindsay Andras, Attending Physician, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-24-00371
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: spinal curve monitoring; Scoliosis mobile application

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Momentum Application (Experimental): Patients diagnosed with scoliosis between 8-18 years of age
  Interventions: Device: Momentum Application

INTERVENTIONS:
Device: Momentum Application — A mobile application to scan and predict spinal curvature. The application monitors curvature and track changes over time.

SUMMARY:
The goal of this clinical trial is for the Momentum SpineTM application to accurately detect scoliosis progression, including accuracy, margin of error, sensitivity, specificity, AUC, and overall agreement with radiographs in 8-18 year olds with adolescent idiopathic scoliosis. The main question it aims to answer [is/are]:

* Based on previous data it is hypothesize that Momentum SpineTM imaging software will be able to accurately detect scoliosis progression (>= 7 degrees), including accuracy, margin of error, sensitivity, specificity, AUC, and overall agreement with radiographs.
* Based on the above hypothesis that Momentum SpineTM is able to accurately detect scoliosis and curve progression (>= 7 degrees).
* It is hypothesized there will be indications for accelerated clinical visits based on at home detection of progression, and that these visits will be accurate and necessary.
* It is hypothesized that there will be a proportion of standard care visits that are deemed unnecessary, and that the application is able to accurately predict these visits.

Participants will:

* Use Momentum SpineTM assessment from home to perform body scans at 1-month intervals on personal device and during the clinical visit.
* Received monthly scans that will be evaluated by the provider using the application.
* Receive additional scans as warranted.
* Complete net promoter score (NPS) within the application following completion of a body scan.
* Complete a patient satisfaction survey following 6 months of application usage.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 8-18 years of age
* Confirmed radiographic diagnosis of adolescent idiopathic scoliosis
* No history of spinal/ chest surgery.
* Participants who have had spine x-rays ±1 week as baseline visit at CHLA will be included in the study.
* Participants who have identifiable markings such as tattoos or birthmarks can be included in the study, though their markings will be covered with tape.

Exclusion Criteria:

* Participants who have had x-rays in a brace will not be included.
* Participants who have had an x-ray from another institution will not be included in the study. X-rays from out of community are typically done with a different and lower quality machine then the one at our institution. Additionally, we do not have consent from outside institutions to use their x-rays for research purposes.
* Participants with a confirmed pregnancy will not be included. Pregnancy status will be self-reported by participants.
* Participants with the existence of a second deformity which may affect topographic assessment will be excluded (e.g. Limb length discrepancy greater than 2cm).
* Families who do not speak English and Spanish will be unable to participate as the application is only available in English and Spanish at this time.
* Families who do not have access to their own compatible personal smart phone device will be unable to participate in the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Scoliosis Progression | Immediately from enrollment and monthly through study completion
  Progression will be defined as a change of greater than or equal to 7 degrees. The progression between the application will be compared to the radiographs done manually, with evaluation of the margin of error, sensitivity, specificity, AUC, and overall agreement with the radiographs.

SECONDARY OUTCOMES:
Proportion of follow-up visits that were correctly accelerated | Immediately from enrollment through study completion, at an average of 2 years
  Accelerated visits are defined as medical appointments less than 6 months apart (sooner than routine follow-up) suggested by the Momentum Spine mobile application. When Momentum Spine detects progression on 3D models obtained at home, it suggests the clinical team see that patient sooner than the planned semi-annual visit in order to implement treatments earlier (bracing, change in brace, etc.). This endpoint will calculate the percentage of accelerated visits suggested by Momentum Spine where scoliosis progression was present as well as where a change in treatment was required.
Necessity of visit | Immediately from enrollment and monthly through study completion
  Coronal curve magnitude between site-specific X-ray measurements and coronal curve magnitude predictions output by Momentum Spine will be compared . The cutoff to determine whether the predicted coronal curve magnitude will be a difference of +/- 7 degrees when compared to the average of the readings from x-rays.
  Progression noted via Momentum Spine and on radiographs will be compared.
  Necessary visit = Radiographic Progression >7 degrees Unnecessary visit = Radiographic Progression <7 degrees
  Percentage agreement between Radiographic and MS progression values, with a cutoff point of 7 degrees, will be assessed.
Proportion of avoidable x-rays using Momentum Spine | Immediately from enrollment and monthly through study completion
  An avoidable x-ray is defined as the percentage of radiographs obtained as part of routine semi-annual follow-up that show an absence of scoliosis progression where Momentum Spine was in agreement. This metric demonstrates that Momentum Spine is an accurate tool for determining when spinal radiographs are necessary.
Patient Satisfaction Survey | Only at the 6 month visit
  The patient satisfaction survey consists of 6 open-ended questions to understand what the experience has been for the individual using the application.
Net Promoter Score | Immediately from enrollment and monthly through study completion
  The Net Promoter Score (NPS) is measured by collecting patient/parent ratings on a 0-10 scale in response to questions on how likely they would use the app. The data is collected via a survey embedded within the product. The score uses a scale between a minimum value of 0 (worst) to a maximum value of 5(best).

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M Andras, MD, Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: No